CLINICAL TRIAL: NCT00908622
Title: Phase II, Blind, Controlled, Randomised Study of the Efficacy of Percutaneous Implantation of Autologous Myoblasts in Patients With Old Infarction
Brief Title: Study of the Efficacy of Percutaneous Implantation of Autologous Myoblasts in Patients With Old Infarction
Acronym: PERCUTANEO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Finabiotech (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIO/REG/PERCUTÁNEO
Record Dates: First submitted 2009-05-25; First posted 2009-05-27 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Old Myocardial Infarction
Keywords: Percutaneous implantation of autologous myoblasts
MeSH Terms: interventions — Cell- and Tissue-Based Therapy; Myocardial Revascularization

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Skeletal myoblasts (Experimental): Percutaneous autologous myoblast implantation
  Interventions: Procedure: Percutaneous autologous myoblast implantation
- No cells (Placebo Comparator): Percutaneous culture medium without cells implantation
  Interventions: Procedure: Cardiac revascularization

INTERVENTIONS:
Procedure: Percutaneous autologous myoblast implantation — Endocavity implantation of autologous myoblasts
  Other Names: Cellular therapy
  Arms: Skeletal myoblasts
Procedure: Cardiac revascularization — Cardiac revascularization
  Arms: No cells

SUMMARY:
The purpose of this study is compare the improvement in global and regional cardiac function measured by echocardiography and magnetic resonance in patients with old myocardial infarction subject to cardiac catheterisation with percutaneous endocavity implantation of autologous myoblasts.

DETAILED DESCRIPTION:
Ischaemic heart disease is one of the main causes of mortality and morbidity. In particular, myocardial infarction (MI) is of special significance, as the heart muscle cannot regenerate so a region's necrosis leads to the formation of a fibrous scar. In the last few years, new treatments have been developed for the acute phase of myocardial infarction.We have managed to slow down disease progression with these new treatments, but it continues to the development of end stage heart failure. This study tries to determine the benefit of cell cardiomyoplasty with autologous myoblasts in patients with old MI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of myocardial infarction, absence of viability.
* Ejection fraction under 40% or 45% in symptomatic patients
* Aged from 30-80 years old.
* Negative pregnancy test (women of childbearing age)
* Informed consent granted

Exclusion Criteria:

* Prior history of tachycardia or ventricular fibrillation (except in the acute phase of MI).
* Myocardial infarction with more than 10 years of evolution.
* Patients positive for HIV, HBV or HCB.
* Patients with organ dysfunction: liver and kidney function
* History of cancer or prior treatment with chemotherapy.
* The patient should not suffer from any concomitant severe and/or uncontrolled medical condition.
* Patients who, due to their geographical, psychiatric or social status, have difficulties in meeting the conditions established in the protocol.
* Pregnant or beast feeding women.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Ejection fraction and wall motion score index measured with M-mode and echocardiography | 12 months after surgery

SECONDARY OUTCOMES:
Wall motion score index measured with echocardigraphy and magnetic resonance in the ITT population | 12 month after surgery
Viability measured with echocardigraphy and magnetic resonance in the ITT population | 12 month after surgery
Incidence of cardiac arrythmias in the ITT population | 12 month after surgery
Ejection fraction measured with echocardiography in the ITT population | 12 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Prósper, MD, Ph.D., Study Director — Clínica Universidad de Navarra
Locations (2):
- Spain (2):
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Clínica Universitaria de Navarra, Pamplona, Navarre